CLINICAL TRIAL: NCT00112658
Title: Randomized Phase II/III Trial Comparing Folririnox Association [Oxaliplatin / Irinotecan / LV5FU2] Versus Gemcitabine in First Line of Chemotherapy in Metastatics Pancreas Cancers Patients
Brief Title: Combination Chemotherapy as First-Line Therapy in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CDR0000430100; FRE-FNCLCC-ACCORD-11/0402; EU-20512
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Gemcitabine; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folfirinox (Experimental)
  Interventions: Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: oxaliplatin
- Gemcitabine (Active Comparator)
  Interventions: Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: fluorouracil
  Arms: Folfirinox
Drug: gemcitabine hydrochloride
  Arms: Gemcitabine
Drug: irinotecan hydrochloride
  Arms: Folfirinox
Drug: leucovorin calcium
  Arms: Folfirinox
Drug: oxaliplatin
  Arms: Folfirinox

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective as first-line therapy in treating pancreatic cancer.

PURPOSE: This randomized phase II/III trial is studying how well combination chemotherapy works as first-line therapy in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the objective response rate in patients with metastatic adenocarcinoma of the pancreas treated with oxaliplatin, irinotecan, leucovorin calcium, and fluorouracil vs gemcitabine as first-line chemotherapy. (Phase II)
* Compare the survival of patients treated with these regimens. (Phase III)

Secondary

* Compare the toxicity of these regimens in these patients.
* Compare progression-free survival of patients treated with these regimens. (Phase III)
* Compare the overall response rate in patients treated with these regimens. (Phase III)
* Compare quality of life of patients treated with these regimens. (Phase III)

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oxaliplatin IV over 2 hours, irinotecan IV over 1½ hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 5 minutes on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Courses repeat every 14 days.
* Arm II: Patients receive gemcitabine IV on days 1, 8, 15, 22, 29, 36, and 43. Beginning on day 57, patients receive gemcitabine IV once weekly for 3 weeks (days 57, 64, and 71). Courses repeat every 28 days.

PROJECTED ACCRUAL: A total of 348 patients (88 for phase II and 260 for phase III) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * No other pancreatic tumor type, including either of the following:

    * Neuroendocrine tumor
    * Acinar cell tumor
  * Metastatic disease
* Measurable disease in an area not previously irradiated
* No cerebral metastases or meningeal involvement of the tumor

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (biliary drainage allowed)

Renal

* Creatinine < 120 mmol/L

Cardiovascular

* No prior myocardial infarction
* No prior angina
* No uncompensated cardiac or coronary insufficiency
* No symptomatic arrhythmia

Gastrointestinal

* No prior inflammatory bowel disease
* No prior chronic diarrhea
* No unresolved symptomatic occlusion or subocclusion of the bowel

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No ongoing active infection
* No other malignancy except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No contraindication to study treatment
* No other serious medical disorder that would preclude study treatment
* No psychiatric disorder or social or geographic situation that would preclude study participation
* Not detained or under the guardianship of another person

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Other

* No concurrent participation in another clinical trial using therapeutic experimental agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (Phase II)
Survival (Phase III)

SECONDARY OUTCOMES:
Toxicity
Progression-free survival (Phase III)
Quality of life (Phase III)
Overall response rate (Phase III)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Conroy, MD, Study Chair — Centre Alexis Vautrin
Locations (55):
- France (55):
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Hopital Duffaut, Avignon
  - Centre Hospitalier General, Belfort
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Avicenne, Bobigny
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - CHU de Caen, Caen
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - CHR Clermont Ferrand, Hotel Dieu, Clermont-Ferrand
  - Hopitaux Civils de Colmar, Colmar
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Hopital Du Bocage, Dijon
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospitalier Intercommunal St. Aubin les Elbeuf, Elbeuf
  - Clinique Saint Vincent, Épernay
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - CMC Les Ormeaux, Le Havre
  - Centre Oscar Lambret, Lille
  - Hopital Saint Vincent de Paul, Lille
  - Polyclinique des Quatre Pavillons, Lormont
  - Hopital de la Croix Rousse, Lyon
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot - Lyon, Lyon
  - Hopital Ambroise Pare, Marseille
  - CHU de la Timone, Marseille
  - CHU Nord, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - Centre Hospitalier General de Mont de Marsan, Mont-de-Marsan
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Saint Michel, Paris
  - Centre Hospitalier de Perpignan, Perpignan
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - CHU - Robert Debre, Reims
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - Clinique Charcot, Sainte-Foy-lès-Lyon
  - Centre Hospitalier de Semur en Auxois, Semur-en-Auxois
  - Centre Paul Strauss, Strasbourg
  - Hopital Universitaire Hautepierre, Strasbourg
  - Centre Hospitalier de Tarbes, Tarbes
  - Institut Claudius Regaud, Toulouse
  - CHU de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Result] Ychou M, Desseigne F, Guimbaud R, et al.: Randomized phase II trial comparing folfirinox (5FU/leucovorin [LV], irinotecan [I] and oxaliplatin [O]) vs gemcitabine (G) as first-line treatment for metastatic pancreatic adenocarcinoma (MPA): first results of the ACCORD 11 trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-4516, 2007.
- [Derived] Lambert A, Jarlier M, Gourgou Bourgade S, Conroy T. Response to FOLFIRINOX by gender in patients with metastatic pancreatic cancer: Results from the PRODIGE 4/ ACCORD 11 randomized trial. PLoS One. 2017 Sep 20;12(9):e0183288. doi: 10.1371/journal.pone.0183288. eCollection 2017. PMID 28931010